CLINICAL TRIAL: NCT05694767
Title: A Prospective, One-arm and Open Clinical Study to Assess Safety and Efficacy of Anti-Human CD38 Monoclonal Antibody CM313 in the Treatment of Primary Immune Thrombocytopenia
Brief Title: A Prospective, One-arm and Open Clinical Study of CM313 in the Treatment of Immune Thrombocytopenia
Acronym: 2022-CM313-ITP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022039（2）
Record Dates: First submitted 2022-12-15; First posted 2023-01-23 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-07

CONDITIONS: Immune Thrombocytopenia; Treatment
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (CM313) (Experimental): 20 enrolled subjects: once a week x 8 doses
  Interventions: Drug: CM313 Injection

INTERVENTIONS:
Drug: CM313 Injection — intravenous CM313 administration
  This study adopts a prospective, single arm, open design method. Twenty subjects were enrolled in the study and were treated with CD38 monoclonal antibody (CM 313: 16mg/kg/w) for 8 weeks.
  The first stage is the main research stage (d1-w8), which is the core treatment period. The subjects will receive intravenous infusion of 16mg/kg CM313 once a week for 8 weeks to observe the safety and efficacy during treatment.
  The second stage (w9-w24) is the stage of withdrawal from the visit, mainly to observe the safety and continuous efficacy of CM313 after treatment.

SUMMARY:
To evaluate the safety and efficacy of CM313 in the treatment of immune thrombocytopenia in patients who have not responded adequately or relapsed after first-line treatment and at least one second-line therapy including rituximab and/or TPO-RA.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an organ-specific autoimmune disease, which is characterized by decreased platelet count and skin and mucosal bleeding. ITP is a kind of disease with increased platelet destruction and impaired platelet production caused by autoimmunity. Conventional treatment of adult ITP includes first-line glucocorticoid and immunoglobulin therapy, second line TPO and TPO receptor agonist, splenectomy and other immunosuppressive treatments (such as rituximab, vincristine, azathioprine, etc.). ITP is one of the most common hemorrhagic diseases. At present, the treatment response of ITP is not good, and a considerable number of patients need drug maintenance treatment, which seriously affects the quality of life of patients and increases the economic burden of patients. Therefore, there is still a lack of effective treatment for adult ITP, especially for recurrent and refractory ITP patients, which is one of the problems that have attracted more attention and need to be solved urgently.

The main pathogenesis of ITP is the loss of platelet autoantigen immune tolerance, which leads to abnormal activation of humoral and cellular immunity. It is characterized by antibody mediated platelet destruction and insufficient platelet production by megakaryocytes. The residual long-term autoreactive plasma cells may be a source of therapeutic resistance to autoimmune cytopenia. Antiplatelet specific plasma cells have been detected in the spleen of patients with rituximab refractory ITP. Therefore, the strategy of simply eliminating B cells may not work, because LLPC will continue to produce pathogenic antibodies. However, targeting LLPC becomes a new strategy to treat autoimmune diseases.

CM313, a kind of anti-CD38 antibody, is a new type of monoclonal antibody targeting CD38. It targets plasma cells and has carried out some clinical studies in multiple myeloma, with good therapeutic effects. In addition, the clinical trials of similar CD38 monoclonal antibody drugs, such as daratumumab, in the treatment of autoimmune diseases, including membranous nephropathy, systemic lupus erythematosus (SLE) and ITP, are also being carried out simultaneously. We assume that autologous reaction LLPC may be the cause of treatment failure in some ITP patients. Therefore, the use of CD38 monoclonal antibody to clear long-term surviving plasma cells in ITP patients may be a new strategy for treating ITP patients.

Therefore, the investigators designed this clinical trial to evaluate the safety and efficacy of CM313 in the treatment of immune thrombocytopenia in patients who are steroid-refractory or steroid-dependent, and fail to respond to at least one previous second-line therapy, including rituximab and/ or TPO agonist.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above, male or female
* Conform to the diagnostic criteria of immune Thrombocytopenia (ITP)
* Diagnosis of ITP ≥3 months, and with a platelet count of <30 X 109/L measured within 2 days prior to inclusion
* Failure to achieve response or relapse after corticosteroid therapy, and at least one second-line therapy including rituximab or TPORAs.
* The previous emergency treatment of ITP (e.g. methylprednisolone, platelet transfusion, IVIG transfusion) must be completed at least 2 weeks before the first administration
* Signed and dated written informed consent
* With normal hepatic and renal functions
* ECOG physical state score ≤ 2 points
* Cardiac function of the New York Society of Cardiac Function ≤ 2
* Patients receiving maintenance treatment (including corticosteroids (less than or equal to 0.5mg/kg prednisone), TPO receptor agonists, etc.) must have a stable dose at least 4 weeks before the first administration, and azathioprine, danazol, cyclosporin A, tacrolimus, sirolimus, etc. must be stopped at least 4 weeks before the first administration; The end of rituximab treatment was>3 months；More than 6 months after splenectomy.

April 10, 2023 After approval by the Ethics Committee on , subjects no longer require platelet glycoprotein autoantibodies positivity upon enrollment.

Exclusion Criteria:

* Received any treatment of anti-CD38 antibody drug
* Uncontrollable primary diseases of important organs, such as malignant tumors, liver failure, heart failure, renal failure and other diseases;
* HIV positive;
* Accompanied by uncontrollable active infection, including hepatitis B, hepatitis C, cytomegalovirus, EB virus and syphilis positive;
* Accompanied by extensive and severe bleeding, such as hemoptysis, upper gastrointestinal hemorrhage, intracranial hemorrhage, etc.;
* At present, there are heart diseases, arrhythmias that need treatment or hypertension that researchers judge is poorly controlled;
* Patients with thrombotic diseases such as pulmonary embolism, thrombosis and atherosclerosis;
* Those who have received allogeneic stem cell transplantation or organ transplantation in the past;
* Patients with mental disorders who cannot normally obtain informed consent and conduct trials and follow-up;
* Patients whose toxic symptoms caused by pre-trial treatment have not disappeared;
* Other serious diseases that may limit the subject's participation in this test (such as diabetes; Severe cardiac insufficiency; Myocardial obstruction or unstable arrhythmia or unstable angina pectoris in recent 6 months; Gastric ulcer, etc.);
* Patients with septicemia or other irregular severe bleeding;
* Patients taking antiplatelet drugs at the same time;
* Pregnant women, suspected pregnancies (positive pregnancy test for human chorionic gonadotropin in urine at screening) and lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-01-22 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy after CM313 treatment within 8 weeks | 8 weeks
  Proportion of subjects with a platelet count ≥ 50 × 10^9/L within 8 weeks after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period
Safety of CM 313 | 24 weeks
  Incidence, severity, and relationship of treatment emergent adverse events after CM 313 treatment

SECONDARY OUTCOMES:
Other efficacy evaluation | 12 weeks
  Including: 1. Proportion of subjects with a platelet count ≥ 50 × 10^9/L at week 2, week 4, week 6，week 8，week 10 and week 12 in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period; 2. Proportion of subjects achieving platelet counts ≥ 50×10^9/L at least once in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the first 12 weeks; 3. Proportion of subjects whose platelet counts ≥ 30×10^9/L and at least two times of baseline platelet count in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids within 8 weeks（two consecutive measurements at least 7 days apart）.
Duration from treatment initiation to platelet count ≥30×10^9/L and ≥50×10^9/L | 12 weeks
  Duration from treatment initiation to platelet count ≥30×10^9/L and ≥50×10^9/L without having received any platelet elevating therapy or having had dose increment of TPO-RA and/or corticosteroids
Cumulative weeks of platelet ≥30×10^9/L and platelet ≥50×10^9/L | 24 weeks
  Cumulative weeks of platelet ≥30×10^9/L and platelet ≥50×10^9/L without having received any platelet elevating therapy or having had dose increment of TPO-RA and/or corticosteroids
Number of subjects with clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale | 24 weeks
  Changes of the subjects' numbers in WHO bleeding score after CM313 treatment according to the reported World Health Organization's Bleeding Scale. The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Measurements of platelet glycoprotein (GP) autoantibodies | 24 weeks
  level of anti-GPIIb/IIIa and Ib/IX antibodies before and after CM313 therapy
Measurements of immunoglobulin quantification | 24 weeks
  The level of IgG, IgA, IgM and IgE quantification before and after CM313 therapy
Measurements of various subsets of immunocompetent cells | 24 weeks
  To assess the changes of the percentage of B cell subsets，regulatory B cells（Breg），regulatory T cells (Treg)，supressor T cells（Ts），monocyte subcets, helper T cells（Th）subsets and the functionally-polarized CD4+ T cell subsets, etc. in peripheral blood mononuclear cells（PBMCs）before and after CM313 therapy, and to compare with the healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months to 36 months after study completion
Access Criteria: Upon request to PI

REFERENCES:
- [Derived] Chen Y, Xu Y, Li H, Sun T, Cao X, Wang Y, Xue F, Liu W, Liu X, Dong H, Fu R, Dai X, Wang W, Ma Y, Song Z, Chi Y, Ju M, Gu W, Pei X, Yang R, Zhang L. A Novel Anti-CD38 Monoclonal Antibody for Treating Immune Thrombocytopenia. N Engl J Med. 2024 Jun 20;390(23):2178-2190. doi: 10.1056/NEJMoa2400409. PMID 38899695